CLINICAL TRIAL: NCT04668300
Title: A Phase II Multi-Arm Study to Test the Efficacy of Oleclumab and Durvalumab in Multiple Sarcoma Subtypes
Brief Title: Oleclumab and Durvalumab for the Treatment of Recurrent, Refractory, or Metastatic Sarcoma
Acronym: DOSa
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0159; NCI-2020-05660 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0159 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2020-08-18; First posted 2020-12-16 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Angiosarcoma; Metastatic Dedifferentiated Liposarcoma; Metastatic Osteosarcoma; Recurrent Angiosarcoma; Recurrent Dedifferentiated Liposarcoma; Recurrent Osteosarcoma; Refractory Dedifferentiated Liposarcoma; Refractory Osteosarcoma
MeSH Terms: conditions — Hemangiosarcoma; Liposarcoma; Osteosarcoma | interventions — durvalumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (oleclumab, durvalumab) (Experimental): Patients receive oleclumab IV over 1 hour every 2 weeks for 5 doses, then every 4 weeks thereafter. Patients also receive durvalumab IV over 1 hour every 4 weeks. Cycle repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Durvalumab; Biological: Oleclumab

INTERVENTIONS:
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Biological: Oleclumab — Given IV
  Other Names: Anti-CD73 Monoclonal Antibody MEDI9447; MEDI9447

SUMMARY:
This phase II trial investigates how well oleclumab and durvalumab work in treating patients with sarcoma that has come back (recurrent) or does not respond to treatment (refractory) or has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as oleclumab and durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the tumor response (Response Evaluation Criteria in Solid Tumors [RECIST]) at 4 months in patients with relapsed/refractory sarcoma. (Cohorts 1 and 2) II. To determine the event-free survival (EFS) rate at 4 months after initiation of the treatment in patients with relapsed/refractory osteosarcoma receiving novel immunotherapeutic agents. (Cohort 3)

SECONDARY OBJECTIVES:

I. To determine the progression-free survival (PFS) rate at 12 weeks after initiation of the treatment in patients with relapsed/refractory sarcoma receiving novel immunotherapeutic agents.

II. To estimate the tumor response (Immune-related Response Criteria [irRC] and RECIST) in patients with relapsed/refractory sarcoma.

III. To evaluate the safety and tolerability of receiving novel immunotherapeutic agents in patients with relapsed/refractory sarcoma.

IV. To estimate the median PFS and overall survival (OS) in patients with relapsed/refractory sarcoma receiving novel immunotherapeutic agents.

EXPLORATORY OBJECTIVES:

I. To determine expression of biomarkers (including but not limited to CD73, PD-1 and PD-L1) in pre & post treatment (tx) samples.

II. Quantification and characterization of the immune infiltrate (and other histologic and immunohistologic changes) from tissue samples prior to treatment initiation and post treatment (biopsy at week 6).

III. Identification/quantification of immunologic changes (CD4+, CD8+, Teff, Treg cells and NK cells) in peripheral blood.

IV. Determining an immunoscore based on baseline tumor sample (identification of molecular response/resistance patterns/future therapy options).

OUTLINE:

Patients receive oleclumab intravenously (IV) over 1 hour every 2 weeks for 5 doses, then every 4 weeks thereafter. Patients also receive durvalumab IV over 1 hour every 4 weeks. Cycle repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years of age or older (cohort 1 and cohort 2); 12 years of age or older (cohort 3)
* Histologically or cytologically confirmed sarcoma that fall into one of the following categories. Patients with low-grade tumors are eligible if there is definite evidence of metastasis or progression

  * Angiosarcoma
  * Dedifferentiated liposarcoma
  * Osteosarcoma
* Must have received and have progressed, are refractory or intolerant to standard therapy appropriate for the specific sarcoma subtype, if there is a standard therapy for the subtype
* Subjects must have at least 1 lesion that is measurable by RECIST

  * A previously irradiated lesion can be considered a target lesion if the lesion is well defined, measurable per RECIST, and has clearly progressed since radiation
  * Subjects undergoing fresh tumor biopsies must have additional non-target lesions that can be biopsied at acceptable risk as judged by the investigator or if no other lesions suitable for biopsy, then a RECIST target lesion used for biopsy must be >= 2 cm in longest diameter
* Subjected must consent to provide archived tumor specimens for correlative biomarker studies. Tumor tissue must be identified and availability confirmed prior to initiation of study therapy. In the setting where archival material is unavailable or unsuitable for use, or there have been multiple intervening therapies subjects must consent and undergo fresh tumor biopsy. A tumor lesion planned for biopsy must not have a RECIST target lesion unless there are no other lesions suitable for biopsy and lesions used for biopsy is >= 2 cm in longest diameter
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (use Karnofsky for patients > 16 years and Lansky for patients =< 16)
* Absolute neutrophil count >= 1.5 x 10^9/L (1,500/mm^3) (without growth factor within 28 days of first dose or transfusion within 14 days of first dose support)
* Platelet count >= 100 x 10^9/L (100,000/mm^3) (without growth factor within 28 days of first dose or transfusion within 14 days of first dose support)
* Hemoglobin >= 9.0 g/dL (without growth factor within 28 days of first dose or transfusion within 14 days of first dose support)
* Calculated creatinine clearance (CrCl) or 24-hour urine CrCl > 40 mL/min Cockcroft-Gault formula (using actual body weight) will be used to calculate CrCl
* Total bilirubin =< 1.5 x upper limit of normal (ULN); for subjects with documented/suspected Gilbert's disease or liver metastases, bilirubin =< 3 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN; for subjects with hepatic metastases, ALT and AST =< 5 x ULN
* Female patients of childbearing potential who are not abstinent and intend to be sexually active with a non-sterilized male partner must use at least 1 highly effective method of contraception (defined below) from the time of screening throughout the total duration of the drug treatment and the drug washout period (90 days after the last dose of durvalumab monotherapy). Non-sterilized male partners of a female patient of childbearing potential must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female patients should also refrain from breastfeeding throughout this period.
* Non-sterilized male patients who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom plus spermicide from the time of screening throughout the total duration of the drug treatment and drug washout period (90 days after the last dose of durvalumab monotherapy). However, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients should refrain from sperm donation throughout this period
* Female partners (of childbearing potential) of male patients must also use a highly effective method of contraception throughout this period as defined below. Notes: Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.
  * Women >= 50 years of age would be considered post-menopausal if they have amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago.

Highly effective methods of contraception, defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly are described below. Note that some contraception methods are not considered highly effective (e.g. male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progesterone-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which is considered highly effective]; and triphasic combined oral contraceptive pills.

* Copper T intrauterine device
* Levonorgestrel-releasing intrauterine system: e.g., Mirena
* Implants: Etonogestrel-releasing implants: e.g. Implanon or Norplant
* Injection: Medroxyprogesterone injection: e.g., Depo-Provera
* Combined pill: Normal and low dose combined oral contraceptive pill
* Patch: Norelgestromin/ethinylestradiol-releasing transdermal system: e.g., Ortho Evra
* Minipill: Progesterone based oral contraceptive pill using desogestrel: Cerazette is currently the only highly effective progesterone-based

  * Life expectancy of at least 6 months
  * Ability to understand the purposes and risk of the study and has signed a written consent form approved by the investigator's Institutional Review Board (IRB)/Ethics Committee
  * Weight >= 35 kg

Exclusion Criteria:

* Prior therapy with anti-PD1, anti-PD-L1 (including durvalumab) or anti-CD73
* Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener syndrome) within the past 2 years. Subjects with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression. Subjects previously treated central nervous system metastases that are radiographically and neurologically stable for at least 28 days and do not require corticosteroids (or any dose) for symptomatic management for at least 14 days prior to first dose of durvalumab and oleclumab are permitted to enroll
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study
* Receipt of any conventional or investigational anticancer therapy within 21 days prior to the first dose of study drug
* Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable. In addition, local treatment (e.g., by local surgery or radiotherapy) of isolated lesions for palliative intent is acceptable beyond the first cycle with prior consultation and in agreement with the principal investigator (PI)
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (e.g., hearing loss) after consultation with the medical monitor
* Current or prior use of immunosuppressive medication within 14 days prior to the first of durvalumab or oleclumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication)
* History of primary immunodeficiency, solid organ transplantation, or previous clinical diagnosis of tuberculosis
* True positive test results for human immunodeficiency virus (HIV) or hepatitis B or hepatitis C
* Receipt of live, attenuated vaccine within 30 days prior to the first dose of investigational products (NOTE: Subjects, if enrolled, should not receive live vaccine during the study and 180 days after the last dose of investigational products)
* Major surgery (as defined by the investigator) within 4 weeks or thoracotomy for pulmonary metastases within 2 weeks prior to first dose of treatment or if still recovering from prior surgery. Local surgery of isolated lesions for palliative intent is acceptable
* Other invasive malignancy, within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) from durvalumab or oleclumab, or compromise the ability of the subject to give written informed consent
* Any condition that, in the opinion of the investigator or sponsor, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Patients with a history of pneumonitis (active within past 6 months) or interstitial lung disease
* Subjects with a history of venous thrombosis within the past 3 months
* Subjects prior history of myocardial infarction, transient ischemic attack, or stroke in the last 3 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Response rate (Cohorts 1 and 2) | At 4 months post treatment initiation
  Defined as complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Event-free survival (Cohort 3) | At 4 months
  Defined as the time from enrollment to disease progression, death, or discontinuation of treatment for any reason (for example toxicity, patient preference, or initiation of new treatment without documented disease progression). Defined by RECIST 1.1. Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analysis of survival data based on the Cox proportional hazards model will be conducted. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure the models are appropriate.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | At 12 weeks
  Defined as the time from treatment onset to either disease progression as defined by RECIST 1.1. Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analysis of survival data based on the Cox proportional hazards model will be conducted. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure the models are appropriate.
Response rate (CR, PR) | Up to 5 years
  Defined by Immune-related Response Criteria (irRC) and RECIST.
Incidence of adverse events (immune-related grade 3 and/or 4 toxicity)per treatment cohort | Up to 5 years
  Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Toxicity data by grade and relationship with the treatment by cohorts and 3 cohorts combined, will be summarized by frequency tables. For the toxicity endpoint, per-treated analysis will be used to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received. Toxicity rate will be estimated with 95% confidence interval.
PFS | Up to 24 weeks
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analysis of survival data based on the Cox proportional hazards model will be conducted. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure the models are appropriate.
Overall survival | Up to 5 years
  Will be estimated using the Kaplan-Meier method. Log-rank test will be performed to test the difference in survival between groups. Regression analysis of survival data based on the Cox proportional hazards model will be conducted. The proportional hazards assumption will be evaluated graphically and analytically, and regression diagnostics (e.g., martingale and Shoenfeld residuals) will be examined to ensure the models are appropriate.

OTHER OUTCOMES:
Biomarker (CD73, PD-1/PD-L1) expression analysis (pre & post treatment tissue samples) | Up to 5 years
  Evaluated using immunohistochemistry (CD73, PD-1/PD-L1) expression analysis). Exploratory data analysis and graphical methods will be applied to examine the distribution of the biomarker data, error checking, and outlier identification. T-test/analysis of variance (ANOVA) or their nonparametric counterparts, Wilcoxon rank-sum test/Kruskal-Wallis test will be used to detect differences of the biomarkers between groups. Linear mixed effect models for repeated measures analysis (Liang, 1986) will be employed to assess the change in biomarkers over time with multi-covariates including disease characteristics (tumor stage, site, pathology), and other prognostic factors. Appropriate transformation of the outcome assessment values will be used to satisfy the normality assumption of linear mixed effect model.
Tumor infiltrating lymphocytes (pre and post treatment tissue samples) | Up to 5 years
  Evaluated using immunofluorescence analysis. Exploratory data analysis and graphical methods will be applied to examine the distribution of the biomarker data, error checking, and outlier identification. T-test/ANOVA or their nonparametric counterparts, Wilcoxon rank-sum test/Kruskal-Wallis test will be used to detect differences of the biomarkers between groups. Linear mixed effect models for repeated measures analysis (Liang, 1986) will be employed to assess the change in biomarkers over time with multi-covariates including disease characteristics (tumor stage, site, pathology), and other prognostic factors. Appropriate transformation of the outcome assessment values will be used to satisfy the normality assumption of linear mixed effect model.
Identification/quantification of immunologic changes (CD4+, CD8+, Teff, Treg cells and NK cells) in peripheral blood | Up to 5 years
  Evaluated using flow cytometry analysis. Exploratory data analysis and graphical methods will be applied to examine the distribution of the biomarker data, error checking, and outlier identification. T-test/ANOVA or their nonparametric counterparts, Wilcoxon rank-sum test/Kruskal-Wallis test will be used to detect differences of the biomarkers between groups. Linear mixed effect models for repeated measures analysis (Liang, 1986) will be employed to assess the change in biomarkers over time with multi-covariates including disease characteristics (tumor stage, site, pathology), and other prognostic factors. Appropriate transformation of the outcome assessment values will be used to satisfy the normality assumption of linear mixed effect model.

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Somaiah, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States